CLINICAL TRIAL: NCT02769325
Title: Atropine in Laparoscopic Gynaecological Surgery (The ALGOS Trial) A Randomised, Double Blind, Controlled Trial
Brief Title: Atropine in Laparoscopic Gynaecological Surgery
Acronym: ALGOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinica Santa Maria (Other)
Responsible Party: Principal Investigator, David Torres, Principal Investigator, Clinica Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSM2016001
Record Dates: First submitted 2016-05-03; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Laparoscopic Surgery; Gynecology
Keywords: atropine; pain, postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Atropine; Sevoflurane; Sugammadex; Ketorolac; Rocuronium; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atropine (Experimental): Patients under a standardised general surgery will receive 1mg atropine (10ml) at induction of anesthesia
  Interventions: Drug: Atropine; Drug: Sevoflurane; Drug: sugammadex; Drug: Ketorolac; Drug: Morphine PCA; Drug: rocuronium; Drug: propofol
- placebo (Placebo Comparator): Patients under a standardised general surgery will receive 10 ml of saline at induction of anesthesia
  Interventions: Drug: Placebo; Drug: Sevoflurane; Drug: sugammadex; Drug: Ketorolac; Drug: Morphine PCA; Drug: rocuronium; Drug: propofol

INTERVENTIONS:
Drug: Atropine — IV atropine 0.1%, 10 ml
  Arms: Atropine
Drug: Placebo — IV saline, 10 ml
  Arms: placebo
Drug: Sevoflurane — All patients will receive anaesthesia based on sevoflurane, titrated to a bis of 45-60
Drug: sugammadex — Patients will receive sugamadex for neuromuscular reversion, if necessary
Drug: Ketorolac — 60 mg IV ketorolac will be administered at induction, and patients will receive 30mg/8h on the postoperative period
Drug: Morphine PCA — Patients will receive a PCA of morphine with a program of 0 (continuous infusion), 1 mg bolus and 8 minutes lockout
Drug: rocuronium — general anaesthesia will use rocuronium 0.6 mg/kg to facilitate intubation
Drug: propofol — for anaesthesia induction, patients will receive 2-3 mg/kg iv propofol

SUMMARY:
This is a double blinded, randomised controlled trial that will compare atropine to placebo for postoperative pain in laparoscopic gynaecological surgery

DETAILED DESCRIPTION:
Patients that meet eligibility criteria will receive a standardised general anesthesia based on sevoflurane and opioids and will be randomised in two groups, using computer generated randomisation system. Allocation concealment is established on opaque envelopes that contain random allocation.

Anesthesia depth will be measured by Bispectral index (BIS), titration of sevoflurane to a BIS of 45-60. In case of neuromuscular block reversal at the end of surgery, sugammadex will be administered.

At induction, 1 mg IV atropine 0.1% OR 10ml saline will be administered, depending on group allocation, on a syringe prepared by an anaesthesiologist not involved in the study.

Patients will receive ketorolac 30 mg/8h, acetaminophen 1g/8h and a morphine IV patient controlled anaesthesia pump (PCA) 0-1-8 Outcomes will be evaluated at the postoperative care unit (PACU) and 24 postoperative hours by an investigator blinded to study group

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) Class I-II, gynaecological laparoscopic surgery lasting ≥30' of laparoscopic time, BMI <35

Exclusion Criteria:

* Known allergies to study drugs, concomitant surgeries, patients with closed angle glaucoma, history of coronary disease or heart insufficiency, beta.blockers

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
24 hours morphine consumption | 24 hours
  morphine consumption, measured 24 post hours, in mg

SECONDARY OUTCOMES:
Pain Visual analog scale at 24 hours | 24 hours
pain visual analog scale at postanesthesia care unit | 2 hours post
number of patients with postoperative nausea and/or vomiting | 24 hours
Patient satisfaction, on a qualitative scale | up to three days
number of patients that refer palpitations | 24 hours
number of patients that refer mouth dryness | 24 hours
number of patients that refer blurred vision | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Santa Maria, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No